CLINICAL TRIAL: NCT03801044
Title: Comparison of Lung Ultrasound and Other Volumetric Methods in Peritoneal Dialysis Patients
Brief Title: Lung Ultrasound in PD Patients
Acronym: LUSiPD
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nuri Baris Hasbal, MD, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 1908
Record Dates: First submitted 2018-12-14; First posted 2019-01-11 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Dialysis; Hypervolemia; VEGF Overexpression
MeSH Terms: conditions — Edema | interventions — Echocardiography; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples for levels of vascular endothelial growth factor and N-terminal pro-brain natriuretic peptide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD patients: All PD patients treated in out unit were enrolled.
  Interventions: Diagnostic Test: NT-BNP, VEGF; Diagnostic Test: Echocardiography; Radiation: Chest Radiography; Diagnostic Test: Lung Ultrasound; Diagnostic Test: Bioelectrical Impedence Analysis

INTERVENTIONS:
Diagnostic Test: NT-BNP, VEGF — VEGF-C levels were measured in the serum samples. R&D Systems kit (Minneapolis, MN) (Catalog Number DVEC00) was used for the assays according to the user instructions. NT-proBNP was measured on the Elecsys 2010 analyzer (Elecsys proBNP Immunoassay; Roche Diagnostics).
Diagnostic Test: Echocardiography — Transthoracic echocardiography was performed by the same cardiologist blinded to all other parameters. It was done while abdomen was empty. LV end diastolic diameter (mm), interventricular septum thickness (mm), posterior wall thickness (mm), ejection fraction (%), left ventricle end diastolic volume (ml), left atrial volume (ml), left ventricle mass index (LVMI) (g/m2), left ventricle filling velocity(cm/sec), E/E' ratio, pulmonary artery systolic pressure (mm Hg) were the parameters taken by echocardiography
Radiation: Chest Radiography — All radiographies were taken when the patient was standing erect position during deep inhalation. They were reported by an expert radiologist blinded to clinical data. Films taken at supine position or during exhalation were excluded. Chest radiographies were classified into 3 stages to reflect degree of hypervolemia. Stage 1 was redistribution defined as increased artery-to-bronchus ratio in the upper and middle lobes. Stage 2 was interstitial edema evident by Kerley B lines and peribronchial cuffing. Stage 3 was alveolar edema phase perihilar consolidation and air bronchograms, pleural fluid, increased width of the vascular pedicle, enlarged cardiac silhouette.
Diagnostic Test: Lung Ultrasound — It was performed by 28 area method which contains ultrasound examination from second to fifth intercostals spaces at parasternal region, midclavicular line, anterior and mid axillary lines. Lung ultrasound had been done by same radiologist who was an expertise in ultrasonography blinded to all other parameters. It was performed by 1,6 megaHertz convex probe when patient lying at the supine position.
Diagnostic Test: Bioelectrical Impedence Analysis — The Body Composition Monitor (BCM) (type 0BJA1394, Fresenius Medical Care AG & Co. KGaA, D-61343 Bad Homburg) was used for assessment of hydration status in patients. Peritoneal cavities were free of intraperitoneal fluid during measurement. Patients were accepted as normovolemic if their result were between -1.1lt and 1.1 lt.

SUMMARY:
Although many alternative methods are present, maintaining ideal volume status in peritoneal dialysis (PD) patients still rely on clinical evaluation due to lack of an evidence based method. Lung ultrasound (LUS) is a new method for evaluation of hidden congestion in this group. LUS findings and its relationship with other volumetric methods are investigated in this study. LUS was performed to all peritoneal dialysis patients and compared with symptoms of hypervolemia, physical examination, vascular endothelial growth factor-C (VEGF-C) and N-terminal pro-brain natriuretic peptide levels, chest radiography, echocardiography, bioelectrical impedance analysis.

DETAILED DESCRIPTION:
Maintaining volume control is crucial in all renal replacement therapy modalities. Fluid overload is associated with increased mortality both in hemodialysis patients and peritoneal dialysis (PD) patients although peritoneal dialysis has the advantage of better preservation of residual renal function compared to hemodialysis. Many methods have been used to fine tune the volume status of patients including physical examination, chest radiography, blood pressure, laboratory parameters, echocardiography, bioelectrical impedance analysis (BIA), ultrasound for lung.

Symptoms of hypervolemia are mainly paroxysmal nocturnal dyspnea, orthopnea, edema, dyspnea on exertion. On physical examination, hypertension or hypotension, third heart sound, jugular venous distension, rales, edema can be seen. Pulmonary venous congestion, cardiomegaly, interstitial edema, alveolar edema, pleural effusion can be seen on chest radiographies.

Level of N-terminal pro-brain natriuretic peptide (NT-proBNP) increases upon stretching of cardiac myocytes. This is accepted as a reflection of volume status. There are a few studies in which NT-proBNP was found as a useful marker for hypervolemia both in hemodialysis and peritoneal dialysis population.

Vascular endothelial growth factor-C (VEGF-C) is an osmosensitive gene product secreted by macrophages through activation of tonicity-responsive enhancer binding protein found in mononuclear phagocyte system cells infiltrating the interstitium. The result is hypertonic sodium accumulation in the skin which is accepted as a buffer mechanism maintaining blood pressure homeostasis. Serum VEGF-C levels had been found as a promising marker of hypervolemia in a hemodialysis patient cohort by a recent study.

Echocardiography has been used extensively in dialysis patients in which a number of parameters have been measured. Bioelectrical impedance analysis (BIA) is another non-invasive bedside method for the evaluation of volume status.

Lung ultrasound (LUS) is a technique that has become popular in nephrology recently. "B lines" or "lung comets" are the reverberation artifacts arising from the pleural line. They are produced due to thickened subpleural interlobular septa by edema.

The gold standard for volume assessment is isotope dilution and neutron activation analysis methods which are only limited to research activities. The best widely accepted, non-invasive, practical, easy to access method has not been decided yet. Moreover evidence is quite scarce for the peritoneal dialysis than hemodialysis or normal renal functioning group. Lung ultrasound is the most recent promising method for volume control.

The investigators aimed to define lung ultrasound findings in our peritoneal dialysis cohort and its relation with other volumetric parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old,
* History of PD more than 3 months,
* Providing written informed consent

Exclusion Criteria:

* Patients younger than 18 years old,
* Unwilling to participate to the study,
* Immobile patients unable to perform test in the same day,
* History of PD less than 3 months,
* Presence of active infection,
* History of lung cancer and/or operations.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All peritoneal dialysis patients in the clinic have been invited to the study. Twenty three patients were enrolled to the study. Two patients excluded from study because of immobility.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Sevinc, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All peritoneal dialysis patients in Sisli Hamidiye Etfal Training and Research Hospital, Nephrology Outpatient Clinic, Istanbul, Turkey have been invited to the study between May and September 2018.
Pre-assignment Details: Total 23 patients accepted to participate in the study, but two of them were excluded because of immobility and not being capable of proceeding with the diagnostic tests
Groups:
- PD Patients: 21 PD patients treated in out unit were enrolled.
  NT-BNP, VEGF: VEGF-C levels were measured in the serum samples. R&D Systems kit (Minneapolis, MN) (Catalog Number DVEC00) was used for the assays according to the user instructions. NT-proBNP was measured on the Elecsys 2010 analyzer (Elecsys proBNP Immunoassay; Roche Diagnostics).
  Echocardiography: Transthoracic echocardiography was performed by the same cardiologist blinded to all other parameters. It was done while abdomen was empty. LV end diastolic diameter (mm), interventricular septum thickness (mm), posterior wall thickness (mm), ejection fraction (%), left ventricle end diastolic volume (ml), left atrial volume (ml), left ventricle mass index (LVMI) (g/m2), left ventricle filling velocity(cm/sec), E/E' ratio, pulmonary artery systolic pressure (mm Hg) were the parameters taken by echocardiography
  Chest Radiography: All radiographies were taken when the patient was standing erect position during deep inhalation. They
Period: Overall Study
Arm/Group | PD Patients
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PD Patients
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 21
Etiology of End-Stage Renal Disease [Count of Participants; unit: Participants]
  Unknown | 12
  Hypertension | 2
  Diabetes Mellitus | 2
  Familial Mediterrenean Fever | 1
  Focal Segmental glomerulosclerosis | 2
  Ig A Nephropathy | 1
  Tuberous Sclerosis | 1
Duration of PD, months [Median (Inter-Quartile Range); unit: Months] | 22 [13 to 49.5]
PD modality, CAPD (%) [Count of Participants; unit: Participants] | 17
Peritoneum Transport Type [Count of Participants; unit: Participants]
  Low | 1
  Low-medium | 10
  High-medium | 7
  High | 3

OUTCOME MEASURES:

1. Primary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Serum VEGF-C Level (pg/ml) by Enzyme-linked Immunosorbent Assay
Description: Assessing the relationship between number of Kerley B lines by ultrasound and serum VEGF-C level (pg/ml) by enzyme-linked immunosorbent assay
Time Frame: 4 months
Population: All peritoneal dialysis patients in the clinic invited to the study. Two patients were excluded because of immobility
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- PD Patients: 21 PD patients treated in out unit were enrolled.
Arm/Group | PD Patients
Number analyzed (Participants) | 21
ng/ml
  All patients | 0.29 [0.23 to 0.34]
  B Line ≤ 1 | 0.25 [0.21 to 0.32]
  B Line > 1 | 0.33 [0.27 to 0.35]
Statistical Analysis 1: Comparison: PD Patients; Test type: Other; p = 0.039, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Dyspnea by Questionnaire
Description: Assessing the relationship between number of Kerley B lines by ultrasound and dyspnea by questionnaire
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Number; unit: percentage of participants
Groups:
- PD Patients: All PD patients except for two patients who were immobile to adhere to diagnostic tests (n=21).
Arm/Group | PD Patients
Number analyzed (Participants) | 21
percentage of participants
  B Lines ≤ 1 | 25
  B lines > 1 | 11.1

3. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Class of New York Heart Association Classification
Description: Assessing the relationship between number of Kerley B lines by ultrasound and class of New York Heart Association Classification
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Number; unit: percentage of NYHA Class 1
Groups:
- PD Patients: All PD patients except two patients who were immobile for adhering to diagnostic tests.
Arm/Group | PD Patients
Number analyzed (Participants) | 21
percentage of NYHA Class 1
  B Lines ≤ 1 | 91.7
  B lines > 1 | 100

4. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Presence of Third Sound/Pretibial Edema by Auscultation/Edema by Physical Examination
Description: Assessing the relationship between number of Kerley B lines by ultrasound and presence of third sound (S3) by auscultation/edema by physical examination
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Count of Participants; unit: Participants
Groups:
- PD Patients: PD patients (n=21)
Arm/Group | PD Patients
Number analyzed (Participants) | 21
Participants
  B Lines ≤ 1 | 0
  B lines > 1 | 0

5. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound Left Ventricle End Diastolic Diameter (mm) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and left ventricle end diastolic diameter (mm) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | PD Patients
Number analyzed (Participants) | 21
cm
  B Lines ≤ 1 | 4.75 [4.12 to 5.25]
  B lines > 1 | 4.3 [4.1 to 4.75]

6. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound Interventricular Septum Thickness (mm) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B by ultrasound and interventricular septum thickness (mm) (mm) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | PD Patients
Number analyzed (Participants) | 21
cm
  B Lines ≤ 1 | 1.0 [0.9 to 1.1]
  B lines > 1 | 1.0 [0.85 to 1.1]

7. Secondary Outcome: Association Between Number of Kerley B by Ultrasound and Posterior Wall Thickness (mm) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B by ultrasound and posterior wall thickness (mm) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | PD Patients
Number analyzed (Participants) | 21
cm
  B Lines ≤ 1 | 1.0 [0.9 to 1.1]
  B lines > 1 | 0.9 [0.85 to 1.05]

8. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Ejection Fraction (%) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and ejection fraction (%) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: percentage of ejection fraction
Arm/Group | PD Patients
Number analyzed (Participants) | 21
percentage of ejection fraction
  B Lines ≤ 1 | 61 [49.7 to 65]
  B lines > 1 | 60 [60 to 62.5]

9. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Left Ventricle End Diastolic Volume (ml) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and left ventricle end diastolic volume (ml) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | PD Patients
Number analyzed (Participants) | 21
ml
  B Lines ≤ 1 | 100 [76.7 to 128.7]
  B lines > 1 | 94 [87.5 to 135]

10. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Left Atrial Volume (ml) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and left atrial volume (ml) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | PD Patients
Number analyzed (Participants) | 21
ml
  B Lines ≤ 1 | 36 [31 to 44.7]
  B lines < 1 | 37 [26 to 41]

11. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Left Ventricle Mass Index (g/m2) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and left ventricle mass index (g/m2) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: g/m2
Arm/Group | PD Patients
Number analyzed (Participants) | 21
g/m2
  B Lines ≤ 1 | 100.5 [70.2 to 129.5]
  B lines > 1 | 75 [69.5 to 92]

12. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Left Ventricle Filling Velocity (cm/Sec) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and left ventricle filling velocity (cm/sec) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: cm/sec
Arm/Group | PD Patients
Number analyzed (Participants) | 21
cm/sec
  B Lines ≤ 1 | 78.5 [56.7 to 86.2]
  B lines > 1 | 74 [65 to 87]

13. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Early Mitral Inflow Velocity and Mitral Annular Early Diastolic Velocity (E/E') Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and early mitral inflow velocity and mitral annular early diastolic velocity (E/E') obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: rate
Arm/Group | PD Patients
Number analyzed (Participants) | 21
rate
  B Lines ≤ 1 | 11.6 [9.8 to 12.6]
  B lines > 1 | 10.7 [9.9 to 11.5]

14. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Pulmonary Artery Systolic Pressure (mmHg) Obtained by the Cardiologist With Echocardiography
Description: Assessing the relationship between number of Kerley B lines by ultrasound and pulmonary artery systolic pressure (mmHg) obtained by the cardiologist with echocardiography
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | PD Patients
Number analyzed (Participants) | 21
mmHg
  B Lines ≤ 1 | 24 [20 to 33.2]
  B lines > 1 | 24 [19 to 29]

15. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and Bioimpedance Analysis [Assessed With the Body Composition Monitor; Normovolemic if Their Result Between -1,1 lt and 1,1 lt)
Description: Assessing the relationship between number of Kerley B lines by ultrasound and bioimpedance analysis [assessed with the body composition monitor; normovolemic if their result between -1,1 lt and 1,1 lt)
Time Frame: 4 months
Population: PD patients (n=21)
Measure: Median (Inter-Quartile Range); unit: liter
Arm/Group | PD Patients
Number analyzed (Participants) | 21
liter
  B Lines ≤ 1 | 0.8 [0.007 to 2.05]
  B lines > 1 | 1.3 [0.1 to 2.1]

16. Secondary Outcome: Association Between Number of Kerley B Lines by Ultrasound and NT-proBNP Level (pg/ml) by Elecsys proBNP Immunoassay
Description: Assessing the relationship between number of Kerley B lines by ultrasound and NT-proBNP level (pg/ml) by Elecsys proBNP Immunoassay
Time Frame: 4 months
Population: PD patients
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | PD Patients
Number analyzed (Participants) | 21
pg/ml
  B Lines ≤ 1 | 3024 [568 to 9397]
  B lines > 1 | 2217 [885 to 3959]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Lung ultrasound is a non-invasive technique, we did not expect any side-effect. And we did not encounter.
Arm/Group | PD Patients
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
The main limitation of this study is a limited number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03801044/Prot_SAP_000.pdf